CLINICAL TRIAL: NCT03885375
Title: Multimodal Imaging Evaluation of Myocardial Involvement in Immunocardiomyopathic Patients
Brief Title: Diagnostic and Imaging Indicators of Immunocardiomyopathic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Immunocardiomyopathy
Record Dates: First submitted 2019-01-02; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-09

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac involvements in autoimmune diseases (AD) is common but underestimated and an early detection remains a clinical challenge for lacking of efficient imaging methods. The objective of the study was to investigate LV myocardial abnormalities in AD patients by multimodal cardiac imaging, including speckle-tracking echocardiology (STE), cardiac magnetic resonance imaging (CMRI) and positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with autoimmune diseases, including systemic lupus erythematosus (SLE), vasculitis, dermatomyositis, sjogren's syndrome, scleroderma, rheumatoid arthritis and IgG4 associated disease.
* Patient is capable of complying with study procedures

Exclusion Criteria:

* Patient is pregnant or nursing
* Patient is complicated with congenital heart disease
* Patient had cardiac surgery before
* Patient is complicated with serious infections
* Patient is complicated with organ failure
* Patient is complicated with tumors
* Patient is diagnosed indefinitely
* Patient has been involved in other clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient is diagnosed with autoimmune diseases, including systemic lupus erythematosus (SLE), vasculitis, dermatomyositis, sjogren's syndrome, scleroderma, rheumatoid arthritis and IgG4 associated disease.
  Patient is capable of complying with study procedures.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in deformational parameters in echocardiography during follow-up period | 6 months - 1 year - 2 years
  global longitudinal strain (%), circumferential strain (%) and radial strain (%) measured by STE in autoimmune diseases
Progression of myocardial fibrosis and edema during follow-up period | 1 year - 2 years
  Late Gadolinium Enhanced, T1 mapping and T2 mapping tested by CMRI
Change in myocardial perfusion during follow-up period | 1 year - 2 years
  SUVmax examined by PET

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hostipal, Beijing, Beijing Municipality, China